CLINICAL TRIAL: NCT03750045
Title: Proposal for Grip Movement Training for Adults With Fine Motor Limitation
Brief Title: Grip Movement Training for Adults With Fine Motor Limitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Terigi Augusto Scardovelli, Principal Investigator, University of Mogi das Cruzes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 56355416.3.0000.5497
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Hand Injuries and Disorders
MeSH Terms: conditions — Hand Injuries; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): For the tests, the volunteers used the access device (Leap Motion) and a computer that were previously installed. The intervention was composed by 8 sessions of 15 minutes each, where the volunteers used a virtual environment attached it to a Leap Motion, which is a sensor that allows to capture the movements that are produced by the hands and reproduce them in a computer through a 3D virtual environment in order to stimulate the execution of their finer movements. The strength (Jamar) and motor coordination (wooden box) evaluations were made in the first, fourth and eighth sessions with the objective of checking the gain progression or not of motion coordination and grip strength.
  Interventions: Diagnostic Test: Jamar; Diagnostic Test: Wooden box; Other: Virtual environment

INTERVENTIONS:
Diagnostic Test: Jamar — The grip strength was evaluated through a dynamometer JAMAR 5030-J, formed by two parallel steel bars, one stationary and a mobile one, which can be adjusted in five different positions. The volunteer was sitting with a neutrally rotated abducted shoulder, elbow flexed at 90°, the forearm in neutral position, and the wrist between 0° and 30° of extension, 0° to 15° of ulnar variance and it was requested that he or she made the grip movement. This test was performed three times with a one-minute-break between each one.
Diagnostic Test: Wooden box — The motor coordination evaluation was made through the measurement of the time spent to perform the task of fitting. To do so, a wooden box was built. In its upper part, there is a circular orifice with 6 cm of diameter.
Other: Virtual environment — The system proposed is composed by a virtual environment and an access device. The Leap Motion was used as the access device, making it possible to capture the movements performed by the hands.

SUMMARY:
This study is to test the system composed by a 3D virtual environment, attached to the Leap Motion, evaluating its effects on the rehabilitation of hand movements in patients with motor alteration.

DETAILED DESCRIPTION:
In order to elaborate the virtual environment, softwares for 3D content creation were used. The virtual environment is formed by four phases, each one having three spheres that are supposed to be inserted, one by one, into a hole located on the scenario floor. Each phase presents a level of difficulty, from pushing the object to performing the grip movement. By the end of each phase, a log file is generated with the time spent on it.

ELIGIBILITY:
Inclusion Criteria:

* men and women with age equal or higher than 18 years old;
* having clinical diagnosis of neurological pathology;
* presenting fine motor coordination deficit and in grip strength;
* being able to understand instructions in order to perform the tasks of the virtual environment;
* minimum score of 23/24 (from a total of 30) in the Mini-Mental State Examination (MMSE)

Exclusion Criteria:

* Not accepting to participate in this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Virtual environment | 120 minutes
  The intervention was composed by 8 sessions of 15 minutes each, where the volunteers used a virtual environment attached it to a Leap Motion, which is a sensor that allows to capture the movements that are produced by the hands and reproduce them in a computer through a 3D virtual environment in order to stimulate the execution of their finer movements.

SECONDARY OUTCOMES:
Wooden box | Immediately after at the Session 1, 4 and 8.
  The motor coordination evaluation was made in the first, fourth and eighth sessions. Each volunteer used three balls, or spheres, of different sizes (small, medium, large). The objective was to insert each ball in each orifice. The time was measured with a chronometer.
Dynamometer JAMAR | Immediately after at the Session 1, 4 and 8.
  The grip strength (kgf) was evaluated in the first, fourth and eighth sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Terigi A Scardovelli, Ph.D, Principal Investigator — University of Mogi das Cruzes
Locations (1):
- Terigi Augusto Scardovelli, Mogi das Cruzes, São Paulo, Brazil